CLINICAL TRIAL: NCT01406392
Title: Sublingual Misoprostol 12,5 mcg Versus Vaginal Misoprostol 25 mcg for Induction of Labour of Alive and Term Fetus : Randomized Controlled Trial
Brief Title: Sublingual Misoprostol for Induction of Labor
Acronym: SUBMISO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Maternidade Escola Assis Chateaubriand (Other)
Responsible Party: Principal Investigator, Daniele Sofia de Moraes Barros Gattas, PhD, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUBMISO
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Labor; Induced
Keywords: Misoprostol; Sublingual; Induced; Labor
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sublingual Misoprostol 12,5mcg (Active Comparator): Sublingual misoprostol or placebo tablete will be administered for each six hours until the maximum dose of 100mcg or eight tablets.
  Interventions: Drug: Sublingual Misoprostol
- Vaginal Misoprostol 25 mcg (Active Comparator): Vaginal misoprostol or placebo tablets will be administered for each six hours until the maximum dose of 200mcg or eight tablets. Each pacient will receve at the same time a sublingual placebo tablet and vaginal misoprostol or sublingual misoprostol and vaginal placebo tablet. It will depend of the randomization.
  Interventions: Drug: Misoprostol 25mcg

INTERVENTIONS:
Drug: Misoprostol 25mcg — Vaginal misoprostol or placebo tablets will be administered for each six hours until the maximum dose of 200mcg or eight tablets.
  Other Names: Prostokos Cytotec
  Arms: Vaginal Misoprostol 25 mcg
Drug: Sublingual Misoprostol — Sublingual misoprostol or placebo tablets will be administered for each six hours until the maximum dose of 100mcg or eight tablets
  Other Names: Prostokos; Cytotec
  Arms: Sublingual Misoprostol 12,5mcg

SUMMARY:
The purpose of this study is to compare effectiveness and safety of a sublingual misoprostol 12,5 mcg with vaginal misoprostol 25 mcg for induction of labour with an alive and term fetus.

DETAILED DESCRIPTION:
Several methods for induction of labour are available. However, the most effective and with less frequency of adverse effects is still unknown. Vaginal misoprostol has been used frequently to induce labour but other routes of administrations have been proposed, such as oral and sublingual. The purpose of this study is to compare effectiveness and safety of sublingual misoprostol 12,5 mcg with vaginal misoprostol 25 mcg administration for induction of labour with an alive and term fetus. A randomized controlled double-blind trial will be carried in two hospitals: Instituto de Medicina Integral Prof. Fernando Figueira and Universidade Federal do Ceará and Instituto de Saúde Elpídio de Almeida, from July 2014 to November 2016. A total of 150 patients must be enrolled. Inclusion criteria are: a) indication for labour induction; b) term pregnancy with alive fetus; Bishop score less than six. Exclusion criteria are: a) previous uterine scar; b) nonvertex presentation; c) non-reassuring fetal status; d) fetal anomalies; e) fetal growth restriction; f) genital bleeding; g) tumors, malformations and/or ulcers of vulva, perineum or vagina. They will be randomized to receive a sublingual misoprostol 12,5 mcg with vaginal placebo tablet or sublingual placebo with vaginal misoprostol 25 mcg tablet. Vaginal tablets will have 25mcg of misoprostol or placebo. Sublingual tablet will have 12,5mcg or placebo. Vaginal misoprostol or placebo tablets will be administered for each six hours until the maximum dose of 200mcg or eight tablets. Primary outcome will be the frequency of tachysystole. Secondary outcomes will be vaginal delivery within 24 hours, hyperstimulation syndrome, cesarean section, severe neonatal morbidity or perinatal death, serious maternal morbidity or maternal death, need of oxytocin for augmentation of labour, number of misoprostol doses needed to bring on labour, interval from first dose to labour and first dose to delivery, failed induction, uterine rupture, need of labour analgesia, instrumental delivery, side effects, maternal death, meconium, non-reassuring fetal heart rate, Apgar scores less than seven at 1st and 5th minutes, admission at neonatal intensive care unit, neonatal encephalopaty, perinatal death and women not satisfied.

ELIGIBILITY:
Inclusion Criteria:

* Indication for labour induction
* Term pregnancy with alive fetus
* Bishop score less than six

Exclusion Criteria:

* Previous uterine scar
* Nonvertex presentation
* Non-reassuring fetal status
* Fetal anomalies
* Fetal growth restriction
* Genital bleeding
* Tumors, malformations and/or ulcers of vulva, perineum or vagina

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Frequency of taquissistoly | 48 hours
  during 48 hours the presence of taquissistoly will be observed

SECONDARY OUTCOMES:
Hyperstimulation Syndrome | 48 hours
  during 48 hours the presence of hyperstimulation syndrome will be observed
changes in the cervix at 12 and 24 hours | 12 and 24 hours
  changes in the cervix
failure to achieve vaginal delivery within 12 and 24 hours | 12 and 24 hours
  failure to achieve vaginal delivery
the mother's preferred route of administration | after 48 hours
  Ask to mother what route of administratios was the best for her
time between the first dose and the onset of labour and delivery | after 48 hours
  to avaluete the time between the first dose and the onset of labour and delivery
duration of labour | after 48 hours
  to avaluete the time of duration of labour
need for oxytocin | after 48 hours
  to avaluete the use of oxytocin during the labour
failed induction of labour | after 48 hours
  to avaluete the faliled induction of labor
Caesarean section and the indications for this procedure | after 48 hours
  to avaluete the number of Caesarean section and the indications for this procedure
need for epidural anaesthesia | after 48 hours
  to avaluete the need for epidural anaesthesia
maternal side effects (nausea, vomiting, diarrhoea, postpartum haemorrhage and fever); | after 48 hours
  to avaluete if occurred any case of maternal side effects (nausea, vomiting, diarrhoea, postpartum haemorrhage and fever);
severe maternal morbidity (uterine rupture, sepsis and admission to intensive care unit) or maternal death | 48 hours
  to avaluete severe maternal morbidity (uterine rupture, sepsis and admission to intensive care unit) or maternal death
meconium in the amniotic fluid | 48 hours
  to avaluete meconium in the amniotic fluid
non-reassuring foetal heart rate | 48 hours
  non-reassuring foetal heart rate
one- and five-minute Apgar scores <7 | after 48 hours
  to avaluete one- and five-minute Apgar scores <7
admission of the newborn to a neonatal intensive care unit | after 48 hours
  to avaluete admission of the newborn to a neonatal intensive care unit
need for neonatal resuscitation | after 48 hours
  to avaluete the need for neonatal resuscitation
severe neonatal morbidity (convulsions and neonatal asphyxiation) or perinatal death. | after 48 hours
  to avaluete severe neonatal morbidity (convulsions and neonatal asphyxiation) or perinatal death.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira (IMIP), Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After publication in scientific journal

REFERENCES:
- [Derived] Gattas DSMB, de Amorim MMR, Feitosa FEL, da Silva-Junior JR, Ribeiro LCG, Souza GFA, Souza ASR. Misoprostol administered sublingually at a dose of 12.5 mug versus vaginally at a dose of 25 mug for the induction of full-term labor: a randomized controlled trial. Reprod Health. 2020 Apr 10;17(1):47. doi: 10.1186/s12978-020-0901-8. PMID 32272959
- [Derived] Gattas DSMB, da Silva Junior JR, Souza ASR, Feitosa FE, de Amorim MMR. Misoprostol administered sublingually at a dose of 12.5 mug versus vaginally at a dose of 25 mug for the induction of full-term labor: a randomized controlled trial protocol. Reprod Health. 2018 Apr 18;15(1):65. doi: 10.1186/s12978-018-0508-5. PMID 29669596